CLINICAL TRIAL: NCT03631446
Title: Drug Use-Results Survey on Picoprep® Combination Powder
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000311
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-10

CONDITIONS: Bowel Cleansing
MeSH Terms: interventions — picosulfate sodium; Magnesium Oxide; Citric Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients administered Picoprep® for bowel cleansing: Patients administered Sodium Picosulfate, Magnesium Oxide and Citric Acid for bowel cleansing
  Interventions: Drug: Sodium Picosulfate, Magnesium Oxide and Citric Acid

INTERVENTIONS:
Drug: Sodium Picosulfate, Magnesium Oxide and Citric Acid — Combination powder for oral solution
  Other Names: Picoprep®

SUMMARY:
The purpose of this survey is to confirm safety and efficacy with patients who are administered the Picoprep® for cleansing of intestinal contents for preparation of colonoscopy and colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients who are administered the Picoprep® for cleansing of intestinal contents for preparation of colonoscopy and colorectal surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being prepared for colonoscopy and colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 1298 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing assessment for colonoscopy | 48 hours after drug administration
  Assessment of each part of large intestine using a bowel cleanliness rating scale
Bowel cleansing assessment for colorectal surgery | 48 hours after drug administration
  Assessment of each part of large intestine using a bowel cleanliness rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational Site (there may be other sites in this country), Shibuya City, Tokyo, Japan